CLINICAL TRIAL: NCT00526851
Title: Oral Cancer Screening: Practices, Knowledge and Opinions of Ohio Nursing Home Dentists
Brief Title: Oral Cancer Screening Among Nursing Home Dentists in Ohio
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE17Z06; P30CA043703 (NIH); CASE17Z06 (Other: Case Comprehensive Cancer Center); CASE-17Z06-CC213
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Head and Neck Cancer
Keywords: lip and oral cavity cancer; oropharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: survey administration — Nursing home dentists practicing in Ohio are contacted through a recruitment letter and are asked to respond to questions regarding oral cancer screening practices, knowledge of oral cancer detection, and opinions about oral cancer screening using a newly developed survey, which is based on parts of an existing, pre-tested instrument (Oral Cancer Prevention and Early Detection Survey).

SUMMARY:
RATIONALE: Learning about oral cancer screening practices, knowledge, and opinions of Ohio nursing home dentists may help the study of oral cancer in the future.

PURPOSE: This clinical trial is studying oral cancer screening among nursing home dentists in Ohio.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop a comprehensive sample of nursing home dentists in Ohio.
* To document knowledge of oral cancer detection among these dentists.
* To describe opinions of these dentists about oral cancer screening competency.
* To describe the current oral cancer screening practices of these dentists.

OUTLINE: Participants are stratified according to geographical location (urban vs rural).

A comprehensive sample of nursing home dentists practicing in Ohio are contacted through a recruitment letter and are asked to respond to questions regarding oral cancer screening practices, knowledge of oral cancer detection, and opinions about oral cancer screening using a newly developed survey, which is based on parts of an existing, pre-tested instrument (Oral Cancer Prevention and Early Detection Survey).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Dentist practicing either full-time or part-time in a nursing home setting in the state of Ohio

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nursing Home Dentists in Ohio
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Knowledge of oral cancer detection among nursing home dentists in Ohio | Cross-Sectional
Opinions of these dentists about oral cancer screening competency | Cross-Sectional
Current oral cancer screening practices of nursing home dentists in Ohio | Cross-Sectional

CONTACTS AND LOCATIONS:
Overall Officials: Suparna A. Mahalaha, DDS, MPH, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States